CLINICAL TRIAL: NCT00099333
Title: An Exploratory Study of the Safety of Substituting Exenatide for Insulin in Patients With Type 2 Diabetes Who Have Been Using Insulin in Combination With Oral Antidiabetic Therapy
Brief Title: Study of the Safety of Substituting Exenatide for Insulin in Patients Using Insulin and Oral Antidiabetic Agents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-MC-GWAK
Record Dates: First submitted 2004-12-10; First posted 2004-12-13 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: exenatide; exendin-4; Amylin; Eli Lilly; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): The subjects will discontinue their insulin and substitute it with exenatide. Subjects will remain on their existing oral diabetic therapy.
  Interventions: Drug: exenatide
- Insulin (Active Comparator): The subjects will remain on their current insulin therapy. Subjects will also remain on their existing oral diabetic therapy.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: exenatide — Exenatide 5 mcg subcutaneously injected twice daily for 4 weeks; then 10 mcg subcutaneously injected twice daily for 12 weeks.
  Other Names: synthetic exendin-4; AC2993; Byetta
  Arms: Exenatide
Drug: Insulin — Insulin will be taken according to the subject's current regimen
  Arms: Insulin

SUMMARY:
This study will look at the safety of substituting exenatide for insulin in patients with type 2 diabetes who are currently taking insulin and oral antidiabetic agent(s).

DETAILED DESCRIPTION:
This is an exploratory, multicenter, open-label, 2-arm, parallel trial. Approximately 30 patients with type 2 diabetes, currently on a sulfonylurea, or meglitinide and/or metformin and insulin therapy, will be randomized to discontinue insulin and substitute it with exenatide or remain on their current diabetes therapy regimen. All patients will continue their current diet and exercise regimen during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients have been treated with insulin for >=3 months up to 12 years.
* HbA1c <=10.5%.
* Body mass index (BMI) between 27 kg/m2 and 40 kg/m2.

Exclusion Criteria:

* Patients previously received exenatide or GLP-1 analogs.
* Patients have been treated for greater than 2 weeks with thiazolidinediones or alpha-glucosidase inhibitors within 3 months prior to screening.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-02; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated hemoglobin) from Baseline to Week 16 | Baseline, Week 16
  Change in HbA1c from Baseline study termination (Week 16)

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - Research Site, Chula Vista, California
  - Research Site, Butte, Montana
  - Research Site, Portland, Oregon
  - Research Site, Nashville, Tennessee
  - Research Site, San Antonio, Texas

REFERENCES:
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356
- [Derived] Davis SN, Johns D, Maggs D, Xu H, Northrup JH, Brodows RG. Exploring the substitution of exenatide for insulin in patients with type 2 diabetes treated with insulin in combination with oral antidiabetes agents. Diabetes Care. 2007 Nov;30(11):2767-72. doi: 10.2337/dc06-2532. Epub 2007 Jun 26. PMID 17595353